CLINICAL TRIAL: NCT05054803
Title: A Phase I/II, Randomized, Double-blind, Placebo-controlled, Parallel, 2-arms Clinical Trial to Assess the Safety and Efficacy of Intrathecal Administration of WJ-MSC in Chronic Traumatic Cervical Incomplete Spinal Cord Injury
Brief Title: Cell Therapy for Chronic Traumatic Cervical Incomplete Spinal Cord Injury
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Banc de Sang i Teixits (Other)
Collaborators: Institut Guttmann (Other); Academic Research Organization (ARO) - VHIR (Unknown); Complexo Hospitalario Universitario de A Coruña (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BST-SCI-02
Record Dates: First submitted 2021-09-14; First posted 2021-09-23 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Spinal Cord Injury Cervical
Keywords: spinal cord injury; Mesenchymal stromal cells; Wharton jelly; Cell therapy
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled, 2-arms, multicenter clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Active treatment and placebo will be released using the same syringe and blinded in a way that it is no possible to distinguish one to the other.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WJ-MSC (XCEL-UMC-BETA) (Experimental): Pre-filled syringe with 4 ± 1 mL containing WJ-MSC in a balanced saline solution supplemented with human albumin.
  Interventions: Drug: WJ-MSC (XCEL-UMC-BETA)
- Placebo (Placebo Comparator): Pre-filled syringe with 4 ± 1 mL containing a balanced saline solution supplemented with human albumin
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: WJ-MSC (XCEL-UMC-BETA) — Administration of 2 Intrathecal infusions of WJ-MSC at day 1 and at 3 months
  Other Names: Tested product
  Arms: WJ-MSC (XCEL-UMC-BETA)
Drug: Placebo — Administration of 2 Intrathecal infusions of placebo at day 1 and at 3 months
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled, multicenter clinical trial in which 18 patients affected with chronic traumatic incomplete cervical spinal cord injury will be randomized to either the active treatment (2 doses of intrathecal WJ-MSC 3 months apart) or to placebo (2 intrathecal infusions, 3 months apart). Thereafter, patients will be followed-up for 12 months for safety and efficacy assessment.

DETAILED DESCRIPTION:
Double-blind, randomized, placebo-controlled, multicenter clinical trial that will include 18 patients affected with chronic traumatic incomplete cervical spinal cord injury who will be randomized 1:1, stratified by center, to one of the 2 treatment arms of the study: WJ-MSC / WJ-MSC (at a dose of 1E6 ± 30% live cells / Kg of weight) or Placebo / placebo. Medication will be administered intrathecally at day 1 and at 3 months. The main objective of the trial is to assess safety at a 12-month follow-up. Secondary objectives include the evaluation of efficacy through clinical response, electrophysiological changes, questionnaires of functionality and quality of life, as well as the presence of anti-HLA antibodies and donor cellularity in the cerebrospinal fluid.

ELIGIBILITY:
Inclusion Criteria:

1. Single spinal cord injury lesion caused by trauma
2. Affected cord segments between C1 and T1, confirmed by magnetic resonance
3. Incomplete lesion (ASIA B, C or D)
4. Chronic disease state (between 1 and 5 years after the injury)
5. Patients from 18 to 70 years of age, both sexes
6. Life expectancy > 2 years
7. Residence near the center during study participation and confidence that the patient will attend the follow-up visits
8. Given informed consent in writing
9. Patient is able to understand the study and its procedures

Exclusion Criteria:

1. Mechanic ventilation
2. Penetrating trauma affecting the spinal cord
3. Pregnant woman or without proper anticonceptive measures according to the investigator, or breath feeding
4. Planned spinal surgery within subsequent 12 month after entering the trial
5. Neurodegenerative diseases
6. Significant abnormal laboratory tests that contraindicates patient's participation in the study
7. Neoplasia within the previous 5 years, or without complete remission
8. Patient with communication difficulties
9. Simultaneous participation in another clinical trial or treated with an investigational medicinal product the previous 30 days, that could interfere in the results of the study
10. Previous treatment with and advanced Therapy Medicinal Product (cell therapy)
11. Contraindication for lumbar punction
12. Contraindication or inability to follow a rehabilitation program
13. Other pathologic conditions or circumstances that difficult participation in the study according to medical criteria
14. The patient does not accept to be followed-up for a period that could exceed the clinical trial length

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | At 12 month follow-up
  Adverse events

SECONDARY OUTCOMES:
American Spinal Injury Association (ASIA) impairment scale | At 1, 3, 4, 6 and 12 month follow-up
  Changes in ASIA score with respect to baseline value as detailed at https://asia-spinalinjury.org/international-standards-neurological-classification-sci-isncsci-worksheet/
Motor evoked potentials | At 6 and 12 month follow-up
  Changes in motor evoked potentials score with respect to baseline value. Higher scores mean a better outcome
Somatosensory evoked potentials | At 6 and 12 month follow-up
  Changes in somatosensory evoked potentials score with respect to baseline value. Higher scores mean a better outcome
Electrical pain threshold perception | At 6 and 12 month follow-up
  Changes in electrical pain threshold perception score with respect to baseline. Lower scores mean a better outcome
Handgrip Strength | At 6 and 12 month follow-up
  Will be assessed using a dynamometer. Changes in the score with respect to baseline values. Higher scores mean a better outcome
Walking index for spinal cord injury (WISCI II) | At 6 and 12 month follow-up
  Changes in the walk test WISCIII score with respect to baseline value. The score ranges from 0 (most severe impairment) to 20 (least severe impairment)
Numerical scale for neuropathic pain assessment | At 6 and 12 month follow-up
  Changes in the numerical scale for neuropathic pain score with respect to baseline value. Score ranges from 0 (no pain) to 10 (unbearable pain)
Modified Ashworth scale for spasticity | At 6 and 12 month follow-up
  Changes in the modified Ashworth scale score with respect to baseline value. It is a 5 point numerical scale that graded spasticity from 0 to 4, with 0 being no resistance and 4 being a limb rigid in flexion or extension, and includes a 1+ value.
Spinal Cord Independence Measure III (SCIM III) | At 6 and 12 month follow-up
  Changes in the SCIM III scale score with respect to baseline value. Score ranges from 0 to 20 with higher scores meaning better outcome.
World Health Organization Quality of life questionnaire (WHOQOL-BREF) | At 6 and 12 month follow-up
  Changes in the WHOQOL-BREF score with respect to baseline value. It contains contains 26 questions each punctuated from 1 to 5 and assesses the individual's overall perception of quality of life (1 to 5), overall perception of their health (1 to 5) and 4 domains of physical health, psychological, social relationships, environment (0-100 each domain). higher scores denote higher quality of life.
Psychological general well-being index (PGWBI) | At 12 month follow-up
  Changes in the PGWBI score with respect to baseline value. Score ranges from 0 to 132, with higher scores meaning a better outcome.
Hospital Anxiety and Depression Scale (HADS) | At 12 month follow-up
  Changes in the HADS score with respect to baseline value. This is a 14-item self-administered questionnaire containing 2 subscales (one for anxiety and one for depression), with a score range of each subscale from 0-21. Higher score indicates higher anxiety and depression.
Community Integration Questionaire (CIQ-IG) | At 12 month follow-up
  Changes in the CIQ-IG score with respect to baseline value. Score ranges from 0 to 25, with higher scores meaning a better outcome.
AntiHLA antibodies in cerebrospinal fluid (CSF) | At 7 days and at 1 month follow-up after each infusion
  Presence or absence of antiHLA antibodies in the CSF after two WJ-MSC infusions
Detection of donor cells in CSF | At 7 days after each infusion
  Short tandem repeat (STR) analysis to detect permanence of donor cellularity (WJ-MsC) in the CSF

CONTACTS AND LOCATIONS:
Overall Officials: Joan VIDAL, MD, PhD, Principal Investigator — Institut Guttmann
Locations (2):
- Spain (2):
  - Hospital de Neurorehabilitació Institut Guttmann, Badalona, Barcelona
  - Complexo Hospitalario Universitario A Coruña (CHUAC), A Coruña

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albu S, Kumru H, Coll R, Vives J, Valles M, Benito-Penalva J, Rodriguez L, Codinach M, Hernandez J, Navarro X, Vidal J. Clinical effects of intrathecal administration of expanded Wharton jelly mesenchymal stromal cells in patients with chronic complete spinal cord injury: a randomized controlled study. Cytotherapy. 2021 Feb;23(2):146-156. doi: 10.1016/j.jcyt.2020.08.008. Epub 2020 Sep 25. PMID 32981857
- See also: Blood and tissue bank of Catalonia, cell producer and sponsor of the trial — https://www.bancsang.net
- See also: Hospital specialized in spinal cord injury — https://www.guttmann.com/
- See also: Hospital specialized in spinal cord injury — https://xxicoruna.sergas.gal/Paxinas/web.aspx?tipo=paxtxt&idContido=595&idLista=4